CLINICAL TRIAL: NCT01525485
Title: Vaginal Electrical Stimulation Versus Sacral Neuromodulation for the Treatment of Refractory Overactive Bladder: A Pilot Study
Brief Title: Vaginal Electrical Stimulation Versus Neuromodulation
Acronym: Estim
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 1104
Record Dates: First submitted 2012-01-19; First posted 2012-02-03 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Refractory Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Electrical Stimulation: Participants will have a dedicated visit with a pelvic floor physical therapist during which instructions on usage and technique for the Minnova unit will be given. The electrical parameters selected will be: 10 Hertz frequency, 5-second on/10=second off cycle, and a pulse width of 0.4 milliseconds. The bipolar square will be delivered over a range that varies from 0 to 100 milliamps, depending on the maximum current intensity comfortably tolerated by the patient. The participant will perform each treatment session for 20 minutes twice daily for 8 weeks. Participants will be asked to keep a log recording the dates, times, and duration of each treatment session.
- Interstim device: Participants assigned to the sacral neuromodulation group will undergo InterStim device placement by one of the three Urogynecologists at OUHSC using a staged implant technique according to manufacturer's specifications.

SUMMARY:
This prospective study compares quality of life measures of patients with refractory overactive bladder, between two modes of neuromodulation: vaginal electrical stimulation (Group A) and sacral nerve stimulation (Group B).

The specific aims are:

1. To characterize patient symptom bother score, quality of life, and body image scores in patients obtaining sacral nerve stimulation, as compared to vaginal electrical stimulation.

- Hypothesis 1: Both modes of neuromodulation will impact patients' scores in quality of life, patient symptoms, and body image questionnaires.

DETAILED DESCRIPTION:
All participants will have a standardized intake history which will include age, weight, history of prior treatment for incontinence, medication list, obstetric and gynecologic history, medical history, and surgical history, as well as a complete review of systems. The physical examination will include vital signs (including BMI), genitourinary exam, including Pelvic Organ Prolapse Quantification (POPQ), and neurologic exam. All patients will undergo spontaneous uroflowmetry, urine dipstick from catheterized specimen, multichannel urodynamics, and 3-day voiding diary. Measurement of post-void residual will also be obtained. Completion of the UDI-69, King's Health Questionnaire10, and the Modified Body Image Perception Scale (MBIS) will also be part of the initial visit 11,12.

All participants taking anticholinergics will undergo a 2 week flush-out period prior to the intake assessment. After the intake assessment, the provider will determine which treatment option is appropriate to the participant, and they will then be assigned to one of the two treatment arms: Group A will use vaginal electrical stimulation using the Empi Intravaginal Stimulation Unit Minnova (Empi, St. Paul, MN, USA) and participants in Group B will receive sacral neuromodulation using InterStim (Medtronic, Minneapolis, MN, USA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory OAB (+/- UUI)*
* Female Gender
* Eligible for both treatment interventions
* Available for 8 weeks of follow-up
* Able to complete study assessments
* Must discontinue anticholinergics within 2 weeks of intervention

Exclusion Criteria:

* Age < 21
* Pregnancy
* Stage 3 or 4 pelvic organ prolapse
* Current use of anticholinergics
* Urinary tract infection
* Undergoing concurrent treatment for pelvic organ prolapse
* Unstable or serious cardiac arrhythmia
* Implanted pacemaker
* Postvoid residual > 100ml
* Unstable seizure disorder
* Dementia or inability to follow instructions

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The projected sample size is 48 patients. We anticipate the recruitment of 16 patients for the InterStim arm of this study and 32 patients who will undergo vaginal electrical stimulation. Participants will be drawn from the University of Oklahoma Urogynecology clinics. Our catchment area includes OU Physicians clinic (private clinic) and Presbyterian Professional Building (resident clinic). Our referral area includes all of Oklahoma as well as the surrounding states. Participants will be recruited by physician referrals as well as by campus advertisements.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Symptom improvement | 3 months
  >50% improvement in symptoms and decrease in frequency of voids and episodes of nocturia. Subjective outcomes will be measured by improvement in scores on the UDI-6, KHG, and MBIS.

CONTACTS AND LOCATIONS:
Overall Officials: S. Abbas Shobeiri, MD, Principal Investigator — Univerisity of Oklahoma Health Sciences Center
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States